CLINICAL TRIAL: NCT01771835
Title: Measurement of Retinal Venous Pressure and Endothelin-1 in Patients With Diabetes Mellitus
Brief Title: Retinal Venous Pressure and ET-1 in Patients With Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 089-CYA-2012
Record Dates: First submitted 2012-10-24; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; retinal venous pressure; endothelin-1
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes patients: Patients with diabetes mellitus type I + II, without diabetic retinopathy

SUMMARY:
Measurement of the circulation in patients with diabetes mellitus and establish a link between retinal venous pressure (RVP) and endothelin (ET-1)levels.

DETAILED DESCRIPTION:
Diabetic retinopathy and maculopathy are the main causes of visual loss. Hyperglycemia as the main risk factor of diabetic retinopathy induced damage to retinal capillaries. These in turn lead to hypoxia in the tissue and promote the release of VEGF (vascular endothelial growth factor) , which in turn increases the vascular pathology. Simultaneously, there is an increased expression of endothelin (ET-1). Endothelin increases vascular tone and regulates the micro-and macro-vascular remodeling.

In ocular blood flow perfusion pressure plays an important role. While in healthy eyes a spontaneous retinal venous pulsation is frequently observed, this is significantly less frequent in diseased eyes. An increased venous pressure lowers the ocular perfusion pressure, and increases the transmural pressure. A measurement of the retinal venous pressure and the hormone ET-1 in the blood will give us a better knowledge of the circulatory changes and their relationship to diabetes.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type I or II
* no diabetic retinopathy

Exclusion Criteria:

* known diabetic retinopathy
* acute or chronic inflammation of the eyes
* narrow angle glaucoma
* minority

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabets mellitus type I or II, without diabetic retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Quantification of retinal venous pressure (RVP) | 30 minutes

SECONDARY OUTCOMES:
Quantification of ET-1 in correlation with RVP | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Josef Flammer, MD, Study Director — University of Basel, Dept. of Ophthalmology
Locations (1):
- University of Basel, Dept. of Ophthalmology, Basel, Switzerland

REFERENCES:
- [Derived] Cybulska-Heinrich AK, Baertschi M, Loesche CC, Schoetzau A, Konieczka K, Josifova T, Flammer J. Patients with diabetic retinopathy have high retinal venous pressure. EPMA J. 2015 Feb 24;6(1):5. doi: 10.1186/s13167-015-0027-1. eCollection 2015. PMID 25793018